CLINICAL TRIAL: NCT06068283
Title: LOTUS: an MHealth Intervention to Improve HIV Prevention Service Engagement Intersectional Stigma Among Racially and Ethnically Diverse Women Who Use Drugs
Brief Title: An MHealth Intervention to Improve HIV Prevention Service Engagement Among Racially Diverse Women Who Use Drugs
Acronym: LOTUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephanie Meyers, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 310548-00001; K01DA055983 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-10-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
Keywords: Stigma; Women; Drug Use; mHealth; HIV Prevention
MeSH Terms: conditions — HIV Infections; Social Stigma

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to either the LOTUS mHealth intervention or an informational control. Participants randomized to the treatment arm will receive access to the LOTUS intervention for 6-months. Participants in the control arm will, in parallel, receive access to an information-only website for 6-months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LOTUS Intervention Arm (Experimental): A mobile, WebApp-based platform to access the LOTUS intervention content.
  Interventions: Behavioral: LOTUS mHealth Intervention Group
- Informational Control Arm (Active Comparator): An information-only website, with content on HIV transmission, PrEP, harm reduction, and resources for women.
  Interventions: Behavioral: LOTUS Control Group

INTERVENTIONS:
Behavioral: LOTUS mHealth Intervention Group — A mobile, WebApp-based intervention comprised of tips for HIV prevention, a community wall for peer interaction and support, HIV prevention monitoring and reminders, guided discussions with a health care professional, a resource database, and a personalized profile. Intervention components are designed to promote HIV prevention service use, reduce stigma and improve social support, coping strategies, and positive affect.
  Arms: LOTUS Intervention Arm
Behavioral: LOTUS Control Group — Access to an information-only website with content on HIV transmission, PrEP, harm reduction, and resources for women.
  Arms: Informational Control Arm

SUMMARY:
The goal of this pilot randomized controlled trial is to assess the feasibility, acceptability, and preliminary impact of the mHeaLth interventiOn To redUce Stigma (LOTUS) intervention to improve HIV prevention service engagement and reduce intersectional stigma among racially diverse women who use drugs. LOTUS is a technology-delivered intervention that provides HIV prevention informational content and tips, peer social support and social networking features, a resource locator, HIV prevention monitoring and reminders (e.g., reminders for HIV/STI testing and PrEP doses), and virtual guided discussions with health care professionals.

DETAILED DESCRIPTION:
The LOTUS intervention is a technology-delivered intervention to improve HIV prevention service engagement and reduce intersectional stigma, guided by the Health Stigma and Discrimination Framework and the Theory of Triadic Influences, for racially and ethnically diverse women who use drugs. LOTUS provides HIV prevention informational content and tips, peer social support and social networking features, a resource locator, HIV prevention monitoring and reminders (e.g., reminders for HIV/STI testing and PrEP doses), and virtual guided discussions with health care professionals. Given the disproportionate HIV-related harms racially and ethnically diverse women who use drugs face, and critical need for HIV prevention mHealth interventions tailored to the unique needs of this population, the current study seeks to accomplish the following aim. The primary aim is to assess the feasibility, acceptability, and preliminary impact of the LOTUS intervention in a pilot randomized controlled trial. Racially and ethnically diverse women who use drugs residing in Southern California (n = 60) will be randomized (2:1) to receive the LOTUS intervention or an informational control for 6-months. The proportion of participants retained, intervention use data, and validated self-reported usability, HIV/STI testing, PrEP use, and intersectional stigma measures will be collected at baseline, 3-, and 6-months to assess LOTUS feasibility, acceptability, and preliminary impact. The investigators hypothesize that participants in the LOTUS intervention will find the intervention to be feasible and usable, and that they will demonstrate significant improvements in HIV prevention service use and intersectional stigma at each follow-up time point when compared to control participants. The investigators will also conduct exit interviews with every other participant randomized to LOTUS (n = 20) to gain feedback on the intervention characteristics, as defined by the Consolidated Framework for Implementation Research, and to elicit suggestions for improvement in anticipation of a future large-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current female identity
* Assigned female at birth
* Report weekly or daily use of opioids and/or stimulants in the past 6 months
* Meet current CDC eligibility criteria for PrEP
* Report low levels of HIV prevention service engagement in the past 6 months
* Not currently, or planning on becoming, pregnant during the study
* Owns a smartphone with internet web-browsing capabilities

Exclusion Criteria:

* 17 years of age or younger
* Current gender identity other than female
* Not assigned female at birth
* Does not report weekly or daily use of opioids and/or stimulants in the past 6 months
* Does not meet current CDC eligibility criteria for PrEP
* Report high levels of HIV prevention service engagement in the past 6 months
* Currently, or planning on becoming, pregnant during the study
* Does not own a smartphone with internet web-browsing capabilities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — To be eligible for participation, participants must report being assigned female at birth and current female identity.
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
LOTUS Feasibility | 6 months
  The feasibility of the LOTUS mHealth intervention will be measured by participant retention and via intervention use data.
LOTUS Acceptability | 6 months
  The acceptability of the LOTUS mHealth intervention will be measured via the System Usability Scale (SUS), with possible scores ranging from 10-50 and higher scores indicating higher acceptability.
HIV Prevention Service Engagement | 6 months
  The percentage of participants who report obtaining an HIV/STI test and/or initiating PrEP

SECONDARY OUTCOMES:
Stigma | 6 months
  Intersectional stigma will be measured via the Intersectional Discrimination Index (InDI), which is comprised of three subscales: anticipated discrimination, day-to-day discrimination, and major discrimination. Anticipated discrimination scores range from 0-4, day-to-day discrimination scores range from 0-18, and major discrimination scores range from 0-13. Higher scores on all subscales indicate higher levels of anticipated or experienced discrimination.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No